CLINICAL TRIAL: NCT00709605
Title: A Phase I, Open Label, CT to Evaluate the Safety, Tolerability and Immunogenicity of a Multiclade Recombinant HIV-1 Adenoviral Vector Vaccine, VRC-HIVADV014-00-VP In Uninfected Adults Randomized to Needle or Biojector Methods of Intramuscular Injection
Brief Title: Phase I Study of HIV Adenoviral Vector Vaccine in Healthy Subjects Using Needle or Biojector Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 080171; 08-I-0171
Record Dates: First submitted 2008-06-28; First posted 2008-07-03 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-05-20

CONDITIONS: HIV Infections
Keywords: HIV Negative; Healthy; Immunity; Preventive; Virus; Healthy Volunteer; HV
MeSH Terms: conditions — HIV Infections; Virus Diseases

INTERVENTIONS:
Drug: VRC-HIVADV014-00-VP

SUMMARY:
This study will compare the immune response and side effects of an experimental HIV vaccine given by two different methods of administration by needle injection or by use of a needle-free device called the Biojector 2000 (Registered Trademark). The vaccine, called VRC-HIVADV014-00-VP, or rAd5, is made using an adenovirus that has been modified to contain DNA that codes for three HIV proteins. It cannot cause HIV or adenoviral infections.

Healthy volunteers who are not infected with the HIV virus may be eligible for this study. Subjects are recruited for two study groups: Group 1 comprises volunteers who are 18 to 50 years old and have never received an HIV vaccine and Group 2 comprises volunteers who are 18 to 55 years old and participated in a prior study in which they received at least one injection of the study rAd5 vaccine.

Subjects in both groups are randomly assigned to receive the vaccine by needle or Biojector 2000 (Registered Trademark) into a muscle in the upper arm. They call a study nurse 2 days after the injection, record their temperature and symptoms on a diary card at home for 5 days after the injection for later review, and visit the clinic two weeks after the injection for a checkup.

The injection is given on the day of enrollment. Additional visits are scheduled at weeks 2, 4, 12 and 24, when subjects are checked for health changes or problems, their use of medications and how they are feeling. Blood samples are collected at all clinic visits. Subjects are tested for HIV at the beginning and end of the study, are asked about their sexual behavior and drug use, and are counseled about HIV risk reduction. Women are tested for pregnancy at the beginning and end of the study.

Participants in Group 2 may undergo apheresis at the 4-week visit. This procedure is done to collect white blood cells for tests to examine the immune response to the vaccine. Blood is collected through a needle in the vein of one arm and directed through a machine that separates the cell components. The white cells are removed and the rest of the blood is returned through the same needle.

Subjects are asked about any social effects they may have experienced from participating in the study. These effects are monitored to make sure participants receive any needed assistance and to learn ways to prevent these problems in the future.

DETAILED DESCRIPTION:
Study Design:

VRC 015 will examine safety, tolerability and immune response to the VRC recombinant adenoviral vector serotype 5 vector vaccine, VRC-HIVADV014-00-VP (rAd5), in uninfected subjects who will be randomized to receive the injection either by needle or Biojector injection. The study will include enrollment of rAd5 vaccine-naive subjects, as well as enrollment of rollover subjects who received at least one rAd5 injection in a prior study that included the rAd5 vaccine. The hypothesis is that the rAd5 vaccine will be safe and immunogenic when administered by either needle or Biojector. The primary objectives are to evaluate the safety and tolerability of the rAd5 vaccine at 10(10) PU dosage in the naive and previously vaccinated, uninfected subjects when administered by needle or Biojectors. The secondary objectives include evaluating the HIV-1-specific humoral and T-cell immune responses and adenovirus serotype 5 (Ad5) antibody responses, and social impacts of participation in an HIV vaccine study. Exploratory evaluations include epitope mapping and other immunogenicity evaluations.

Product Description:

The VRC HIV rAd5 vaccine is a recombinant product composed of 4 adenoviral vectors (in a 3:1:1:1 ratio) that encode the HIV-1 Gag/Pol polyprotein from clade B and HIV-1 Env glycoproteins from clades A, B, and C, respectively.

Subjects:

Group 1 will include healthy adults, ages 18-50 years old who are HIV vaccine-naive. Group 2 will include healthy adults, ages 18-55 years old, who are rollover enrollments from a prior study of the VRC HIV rAd5 vaccine.

Study Plan:

Study Group 1 and Group 2 will be simultaneously enrolled. Both groups will be randomized in 1:1 ratio to receive the study injection by needle or Biojector. All study injections will be at a dosage of 10(10) particle units (PU) of rAd5 vaccine delivered into deltoid muscle.

There are more than 100 past study participants who are potentially eligible for Group 2. The study design is based on at least 10 rollover subjects, but allows for additional rollover enrollment of up to 10 more (i.e., Group 2 total n=20) if there is greater than expected interest in participation. The sample for immunogenicity studies collected at Week 4 after vaccination from Group 2 subjects will be obtained by apheresis from those who are willing and eligible for apheresis; otherwise peripheral blood mononuclear cells (PBMCs) will be obtained from 80 mL blood collected by phlebotomy.

Study Duration:

Subjects will be evaluated at 5 or more clinical visits for 24 weeks after the study injection and then followed by annual clinic telephone or mail contact for the subsequent 4 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

1. 18 to 50 years old if enrolling into Group 1 or 18 to 55 years old if enrolling into Group 2.
2. HIV vaccine naive if enrolling into Group 1, or receipt of the VRC HIV rAd5 vaccine in a previous study without experiencing a serious adverse event attributed (i.e., definitely, probably, possibly, or probably not related) to the vaccine if enrolling into Group 2.
3. Available for clinical follow-up through Week 24 of the study and committed to four years of annual follow-up contact after Week 24.
4. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
5. Complete an Assessment of Understanding that includes understanding of the STEP Study results prior to enrollment and verbalize understanding of all questions answered incorrectly.
6. Able and willing to complete the informed consent process.
7. Willing to receive HIV test results and willing to abide by NIH guidelines for partner notification of positive HIV results.
8. Willing to donate blood for sample storage to be used for future research.
9. Willing to discuss HIV infection risks, amenable to risk reduction counseling, committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit, and assessed by the clinic staff as being at low risk of HIV infection on the basis of behaviors in the 12 months before enrollment as follows:

   * Sexually abstinent OR
   * Had two or fewer mutually monogamous relationships with partners believed to be HIV-uninfected and who did not use injection drugs, crack cocaine or methamphetamine OR
   * Had two or fewer partners believed to be HIV-uninfected and who did not use injection drugs, crack cocaine or methamphetamine and with whom he/she regularly used condoms for vaginal or anal intercourse.
10. In good general health without clinically significant medical history.
11. Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) less than or equal to 40 within the 56 days prior to enrollment.

    Laboratory Criteria within 56 days prior to enrollment:
12. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.0 g/dL for men.
13. White blood cells (WBC) = 3,300-12,000 cells/mm(3).
14. Differential either within institutional normal range or accompanied by site physician approval.
15. Total lymphocyte count greater than or equal to 800 cells/mm(3).
16. Alanine aminotransferase (ALT) less than or equal to 1.25 times the upper limit of normal
17. Serum creatinine less than or equal to 1 time the upper limit of normal (less than or equal to 1.3 mg/dL for females; less than or equal to 1.4 mg/dL for males).
18. HIV-uninfected as evidenced by a negative FDA-approved HIV diagnostic blood test if enrolling into Group 1 or negative HIV polymerase chain reaction (PCR) test if enrolling into Group 2
19. Negative hepatitis B surface antigen (HbsAg).
20. Negative anti-HCV (hepatitis C virus antibody) and negative HCV PCR.

    Female-Specific Criteria:
21. Negative beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.
22. A female participant must meet any of the following criteria:

No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

or

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 24 of the study,

or

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 24 of the study by one of the following methods:

* condoms, male or female, with or without a spermicide
* diaphragm or cervical cap with spermicide
* intrauterine device
* contraceptive pills or patch, Depo-Provera or other FDA-approved contraceptive method
* male partner has previously undergone a vasectomy.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

Women:

1. Woman who is breast-feeding or planning to become pregnant during the 24 weeks of study participation.

   Volunteer has received any of the following substances:
2. Immunosuppressive medications, cytotoxic medications, inhaled corticosteroids, or long-acting beta-agonists within the past three months.

   [Note: The following will NOT exclude study participation:
   * use of corticosteroid nasal spray for rhinitis;
   * topical corticosteroids for an acute uncomplicated dermatitis;
   * short-acting beta-agonists in controlled asthmatics; a short course (10 days or less) of corticosteroids for a non-chronic condition completed at least 2 weeks prior to enrollment in this study]
3. Blood products within 112 days (16 weeks) prior to HIV screening.
4. Immunoglobulin within 56 days (8 weeks) prior to HIV screening.
5. Investigational research agents within 28 days (4 weeks) prior to initial study vaccine administration.
6. Live attenuated vaccines within 28 days (4 weeks) prior to initial study vaccine administration.
7. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days (2 weeks) prior to study vaccine administration.
8. Current anti-tuberculosis prophylaxis or therapy.

   Volunteer has a history of any of the following clinically significant conditions:
9. Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain.
10. Autoimmune disease or immunodeficiency.
11. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.
12. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
13. Thyroid disease that is not well-controlled
14. A history of hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
15. Generalized idiopathic urticaria within the last 1 years.
16. Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.
17. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
18. Within the 12 months prior to enrollment: newly-acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2, chlamydia, pelvic inflammatory disease, trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B.
19. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
20. Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizure that have not required treatment within the last 3 years.
21. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
22. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within five years prior to enrollment, history of a suicide plan or attempt.
23. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent.
24. Within the 12 months prior to enrollment, one or more of the following:

    * excessive daily alcohol use
    * frequent binge drinking
    * chronic marijuana abuse
    * any other illicit drug use

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2008-06-25; Primary Completion 2014-05-20 (Actual); Study Completion 2014-05-20 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity, lab tests, AEs)

SECONDARY OUTCOMES:
Immunogenicity (cellular and humoral immune function assays)

CONTACTS AND LOCATIONS:
Overall Officials: Barney S Graham, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Osmanov S, Pattou C, Walker N, Schwardlander B, Esparza J; WHO-UNAIDS Network for HIV Isolation and Characterization. Estimated global distribution and regional spread of HIV-1 genetic subtypes in the year 2000. J Acquir Immune Defic Syndr. 2002 Feb 1;29(2):184-90. doi: 10.1097/00042560-200202010-00013. PMID 11832690
- [Background] Hemelaar J, Gouws E, Ghys PD, Osmanov S. Global and regional distribution of HIV-1 genetic subtypes and recombinants in 2004. AIDS. 2006 Oct 24;20(16):W13-23. doi: 10.1097/01.aids.0000247564.73009.bc. PMID 17053344
- [Background] Catanzaro AT, Koup RA, Roederer M, Bailer RT, Enama ME, Moodie Z, Gu L, Martin JE, Novik L, Chakrabarti BK, Butman BT, Gall JG, King CR, Andrews CA, Sheets R, Gomez PL, Mascola JR, Nabel GJ, Graham BS; Vaccine Research Center 006 Study Team. Phase 1 safety and immunogenicity evaluation of a multiclade HIV-1 candidate vaccine delivered by a replication-defective recombinant adenovirus vector. J Infect Dis. 2006 Dec 15;194(12):1638-49. doi: 10.1086/509258. Epub 2006 Nov 8. PMID 17109335
- [Derived] Sarwar UN, Novik L, Enama ME, Plummer SA, Koup RA, Nason MC, Bailer RT, McDermott AB, Roederer M, Mascola JR, Ledgerwood JE, Graham BS; VRC 015 study team. Homologous boosting with adenoviral serotype 5 HIV vaccine (rAd5) vector can boost antibody responses despite preexisting vector-specific immunity in a randomized phase I clinical trial. PLoS One. 2014 Sep 29;9(9):e106240. doi: 10.1371/journal.pone.0106240. eCollection 2014. PMID 25264782